CLINICAL TRIAL: NCT04556214
Title: Liver Transplantation for Non-Resectable Intrahepatic Cholangiocarcinoma: a Prospective Exploratory Trial (TESLA Trial)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Oslo University Hospital (Other)
Responsible Party: Principal Investigator, Magnus Smedman, MD, Consultant, gastrointestinal oncology, Oslo University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: TESLA trial
Record Dates: First submitted 2020-06-30; First posted 2020-09-21 (Actual); Last update posted 2023-04-11 (Actual); Status verified 2023-04

CONDITIONS: Intrahepatic Cholangiocarcinoma
MeSH Terms: conditions — Cholangiocarcinoma | interventions — Liver Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Liver Transplant (Experimental): The patients will be transplanted according to standard procedures by the institutional protocol. The transplantation procedure is initiated by an exploratory laparotomy with clinical assessment and frozen section of the lymphnodes in the hepatoduodenal ligament and along the common hepatic artery/coeliac axis. Evidence of disease dissemination to these regional lymph nodes will be an absolute contraindication to transplantation.
  Interventions: Procedure: Liver Transplant

INTERVENTIONS:
Procedure: Liver Transplant — Liver Transplant

SUMMARY:
The study will investigate whether liver transplantation provides increased survival, low side effects and good quality of life in patients with bile duct cancer where the tumor cannot be removed by normal surgery. Analyzes of blood and tissue samples from the tumor will be investigated to see if the analyzes can indicate who may have recurrence of the disease after liver transplantation. Furthermore, the effect of chemotherapy on normal liver and tumor tissues in the liver that are removed during transplantation will be investigated..

ELIGIBILITY:
Inclusion Criteria:

* Histologically verified diagnosis of Intrahepatic Cholangiocarcinoma (iCCA)
* First time iCCA or liver only recurrence after previous liver resection for iCCA
* Disease deemed not eligible for liver resection based on tumor location or underlying liver dysfunction
* No vascular invasion, extrahepatic disease, or lymph node involvement detected on imaging
* No signs of extrahepatic metastatic disease according to positron emission computed tomography (PET-CT) scan
* Patient must be accepted for transplantation before progressive disease on chemotherapy.
* Twelve months or more time span from the diagnosis of iCCA and date of being listed for liver transplantation
* No signs of extrahepatic metastatic disease according to CT or magnetic resonance (MR) scan within 4 weeks prior to the faculty meeting at the transplant unit
* At least 18 years of age
* Good performance status, Eastern Cooperative Oncology Group (ECOG) 0 or 1
* Signed informed consent and expected cooperation of the patients for the treatment and follow up
* Received at least 6 months of chemotherapy or locoregional therapy

Exclusion Criteria:

* Major vascular involvement of the tumor
* Perforation of the visceral peritoneum
* Weight loss >15% the last 6 months
* Patient BMI > 30
* Other malignancies, except curatively treated more than 5 years ago without relapse
* Known history of human immunodeficiency virus (HIV) infection
* Prior history of solid organ or bone marrow transplantation
* Substance abuse, medical, psychological, or social conditions that may interfere with the patient's participation in the study or evaluation of the study results
* Known hypersensitivity to rapamycin
* Prior extrahepatic metastatic disease
* Women who are pregnant or breast feeding
* Any reason why, in the opinion of the investigator, the patient should not participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2020-06-01 (Actual); Primary Completion 2035-05-31 (Estimated); Study Completion 2035-05-31 (Estimated)

PRIMARY OUTCOMES:
Overall Survival (OS) | From screening and until 36 months after inclusion
  OS as assessed by quality of life questionnaire (QLQ-C30) patient reported outcome

SECONDARY OUTCOMES:
Overall Survival from time of relapse | From time of relapse and until 36 months after inclusion
  OS as assessed by QLQ-C30 patient reported outcome
Disease free survival | After liver transplantation and up 10 years after liver transplantation
  CT-scan/MRI scan according to RECISTcriteria
Start of new treatment/Change of strategy | Immediately after liver transplatation to start of new treatment
  Time to start of new treatment
Time to decrease in physical function and global health score | Up to 10 years after liver transplantation
  Quality of life measured by EORTC QLQ-C30),
Liver transplant Complication | Up to 90 days after liver transplantation
  Number of Clavien-Dindo grad 3-5 complications
Number of Participants Developing other Malignancies | Up to 10 years after liver transplantation
  Diagnosis of other malignancies
Survival in relation to biological markers | After Liver Transplant until 10 years after liver transplantation
  CEA, CA 19-9 and Germline DNA analyses

CONTACTS AND LOCATIONS:
Overall Officials: Magnus Smedman, MD, Principal Investigator — Oslo University Hospital; Sheraz Yaqub, MD, PhD, Principal Investigator — Oslo University Hospital
Locations (1):
- Oslo University Hospital, Oslo, Norway

REFERENCES:
- [Derived] Achurra P, Fernandes E, O'Kane G, Grant R, Cattral M, Sapisochin G. Liver transplantation for intrahepatic cholangiocarcinoma: who, when and how. Curr Opin Organ Transplant. 2024 Apr 1;29(2):161-171. doi: 10.1097/MOT.0000000000001136. Epub 2024 Jan 23. PMID 38258823